CLINICAL TRIAL: NCT03964064
Title: 3D-printing Template-assisted CT-guided I125 Seed Implantation and Stereotactic Radiotherapy for Locally Advanced Pancreatic Cancer:A Prospective Multicenter Cohort Study
Brief Title: I125 Seed Implantation vs Stereotactic Radiotherapy for Pancreatic Cancer
Acronym: Ckvssip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing 302 Hospital (Other); Guangxi Ruikang Hospital (Other); Tengzhou Central People's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BYSY-CKSI-PC
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Pancreatic Cancer Non-resectable; Brachytherapy; Radiotherapy
Keywords: Pancreatic Cancer Non-resectable; I125 seed implantation; Stereotactic radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- I125 Seed Implantation (Experimental): 3D-printing Template-assisted CT-guided I125 Seed Implantation Prescription dose: gtv140-160gy ctv100-140gy Particle activity: 0.4-0.5mCi
  Interventions: Radiation: Stereotactic Radiotherapy
- Stereotactic Radiotherapy (Experimental): According to the tumor volume, location, organ function and other factors, the dosage of stereotactic directional radiotherapy was determined. The range of BED value of radiotherapy was 80-100 for tumors above 5 mm from gastrointestinal tract and 60-80 for tumors below 5 mm from gastrointestinal tract.
  Interventions: Radiation: 3D-printing Template-assisted CT-guided I125 Seed Implantation

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy — GTV: Combining localization and fusion images to delineate the tumors seen PTV = GTV + 0-10mm Target volume radiation dose: The range of BED value of radiotherapy was 80-100 when the distance between the tumor and gastrointestinal tract was more than 5 mm (alpha/beta=10) and 60-80 when the distance between the tumor and gastrointestinal tract was less than 5 mm (alpha/beta=10).
  Normal Tissue Limit: Reference to TG101 Report
  Arms: I125 Seed Implantation
Radiation: 3D-printing Template-assisted CT-guided I125 Seed Implantation — CT-guided radioactive 125I particle therapy with 3D printing template for pancreatic cancer Preoperative planning Design and fabrication of 3D-PNCT Particle implantation Postoperative dose assessment: CT scan was performed after operation, and the image was transmitted to BTPS for dose verification . The dosimetric parameters included tumor volume, D90, mPD, V100, V150 and V200.
  Arms: Stereotactic Radiotherapy

SUMMARY:
Data of 100 patients with locally advanced pancreatic cancer who received stereotactic radiotherapy or ct-guided radioactive 125I seed implantation in the multicenter of the research group from July 2019 to June 2021 were collected, as well as follow-up data.To evaluate the clinical efficacy of stereotactic radiotherapy and ct-guided 125I seed therapy with 3D printing template in pancreatic cancer;In addition, the local control rate and side effects of ct-guided radioactive 125I particles in the treatment of pancreatic cancer lesions were explored, and the efficacy and safety of different doses of stereotactic radiotherapy were determined.

DETAILED DESCRIPTION:
1. Radiation: Stereotactic Radiotherapy 1.1 Equipment: Accuray VSI Cyberknife stereotactic radiotherapy platform, simulated positioning CT machine, MR, positron emission computed tomography PET-CT, vacuum pad.

   1.2 Radiotherapy localization: CT, MRI and PETCT were used to simulate localization.

   1.3 Relevant Definitions of Tumor Targets CT, MRI, PET-CT fusion, combined with MRI location and PET-CT location image for sketching.

   To delineate target areas and organs at risk. GTV: Combining localization and fusion images to delineate the tumors seen PTV = GTV + 0-10mm Dangerous organs: The stomach, duodenum, jejunum, ileum, colon, spinal cord and esophagus were delineated on the base sequence of CT plain scan.

   The target area should be approved by at least one physician in charge or by a physician in charge.

   1.4 Target volume radiation dose: According to the volume, location, organ function and other factors, the dosage of radiotherapy was determined. The range of BED value of radiotherapy was 80-100 when the distance between the tumor and gastrointestinal tract was more than 5 mm (alpha/beta=10) and 60-80 when the distance between the tumor and gastrointestinal tract was less than 5 mm (alpha/beta=10).

   1.5 Normal Tissue Limit: Reference to TG101 Report
2. CT-guided radioactive 125I seeds therapy with 3D printing template for pancreatic cancer 2.1 Preoperative planning 2.2 Design and fabrication of 3D-PNCT 2.3 125I seeds implantation: 3D-PNCT was placed on the surface of the patient's treatment area, and positioned with the help of the patient's outline features, laser lines, body surface positioning lines and template alignment reference lines.

The location of the template and the tumor is well repeated. If there are errors, the template should be adjusted in time. The insertion needle was percutaneously punctured to a predetermined depth through a template guide hole. During the puncture process, the puncture path was monitored by CT scanning and fine-tuned if necessary to avoid injuring nerves and blood vessels. Seeds implantation and CT scan were performed according to the preoperative plan to understand the distribution of seeds. During the operation, the implant needle should be added or reduced when necessary to ensure that the whole target area is adequately irradiated and the surrounding normal tissues are protected.

2.4 Postoperative dose assessment: CT scan was performed after operation, and the image was transmitted to BTPS for dose verification (Figure 3-4). The dosimetric parameters included tumor volume, D90, mPD, V100, V150 and V200.

After these treatments,to evaluate the clinical efficacy of stereotactic radiotherapy and ct-guided 125I seed therapy with 3D printing template in pancreatic cancer;In addition, the local control rate and side effects of ct-guided radioactive 125I particles in the treatment of pancreatic cancer lesions were explored, and the efficacy and safety of different doses of stereotactic radiotherapy were determined.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old;
* Pathologically diagnosed pancreatic cancer patients;Follow-up treatment is in accordance with the NCCN2019 guidelines for standard treatment.
* Clinical MDT discussion, for the unresectable locally advanced pancreatic cancer, AJCC version 8 pancreatic cancer stage T4N0M0

Arterial invasion:

The pancreatic head and neck tumor invasion of pancreas superior mesenteric artery exceed 180 °;More than 180 ° celiac tumor invasion;The tumor invaded the first jejunal branch of the superior mesenteric artery.The pancreatic body tail superior mesenteric artery or celiac tumor invasion more than 180 °;The tumor invaded the abdominal trunk and abdominal aorta.

Venous invasion:

Tumor invasion or embolization (tumor thrombus or thrombus) of the head and neck of the pancreas leads to unresectable superior mesenteric vein or portal vein reconstruction;The tumor invaded the proximal end jejunal drainage branch of most superior mesenteric veins.The invasion or embolization of a tumor in the tail of the pancreas (thrombus or thrombus) leads to the unresectable reconstruction of the superior mesenteric vein or portal vein.

* ECOG physical condition score: 0-1, Karnofsky score 60, able to withstand puncture;
* Expected survival 3 months;
* Good function of main organs, no severe hypertension, diabetes and heart disease.
* Signed informed consent;
* Has a good compliance, families agree to accept the survival follow-up.

Exclusion Criteria:

* Non-locally advanced pancreatic cancer.
* Participated in other drug clinical trials within four weeks;There was a history of bleeding, and any bleeding event with severe grade of CTCAE5.0 or above occurred within 4 weeks before screening;
* Screening of patients with known central nervous system metastasis or a history of central nervous system metastasis.
* Patients with hypertension who cannot obtain good control by single antihypertensive drug treatment (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg);Having a history of unstable angina pectoris;Patients newly diagnosed with angina within 3 months before screening or myocardial infarction within 6 months before screening;Arrhythmia (including QTcF: 450ms in male and 470ms in female) requires long-term use of anti-arrhythmia drugs and New York heart association grade II cardiac dysfunction;
* Long-term unhealed wounds or incomplete fracture healing;
* Imaging showed that the tumor had invaded important blood vessels or the researchers judged that the patient's tumor had a very high possibility to invade important blood vessels during the treatment and cause fatal bleeding;
* Coagulation function abnormalities, have bleeding tendency;Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues;The use of low-dose warfarin (1mg oral, once daily) or low-dose aspirin (no more than 100mg daily) for preventive purposes is permitted on the premise that the international standardized ratio of prothrombin time (INR) is 1.5;
* Screening for the occurrence of hyperactive/venous thrombosis events in the first 6 months, such as cerebrovascular accidents (including temporary ischemic attack), deep vein thrombosis (except for venous thrombosis caused by intravenous catheterization in the early stage of chemotherapy, which was determined by the researchers to have recovered) and pulmonary embolism, etc.
* Thyroid function was abnormal in the past and could not be kept within the normal range even in the case of drug treatment.
* Attending has a history of psychotropic drug abuse, and can't attend or has mental disorder;
* Always half a year after abdominal tumor lesion radiation;
* Immunodeficiency disease, or has other acquired, congenital immunodeficiency disease, or has a history of organ transplantation;
* Judgment according to the researchers, there is serious to endanger the safety of patients or patients completed the research associated with disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 3 years after the treatment
  The time from enrollment to death from any cause
Progression-free survival (PFS) | 3 years after the treatment
  the time interval of disease progression since the date of diagnosis

SECONDARY OUTCOMES:
Local control rate，LCR | 3 years after the treatment
  patients free from the disease in neck during the follow-up time
Pain score | 1 years after the treatment
  The pain relief of patients before and after treatment was evaluated by digital scoring method
Qol: Quality of Life Score of Tumor Patients | 3 years after the treatment
  Quality of Life Score of Tumor Patients
Adverse reactions | 1 years after the treatment
  Adverse reactions during and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, Chairman, Study Chair — Peking University Third Hospital; Fei Xu, Principal Investigator — Peking University Third Hospital; Xuezhang Duan, Director, Study Director — Beijing 302 Hospital; Kaixian Zhang, Director, Study Director — Tengzhou Central People's Hospital; Zuping Lian, Director, Study Director — Guangxi Ruikang Hospital; Zhe Ji, Study Director — Peking University Third Hospital; Jing Sun, Study Director — Beijing 302 Hospital
Locations (4):
- China (4):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The fifth medical center of PLA general hospital, Beijing, Beijing Municipality
  - Guangxi Ruikang Hospital, Nanning, Guangxi
  - Tengzhou Central People's Hospital, Tengzhou, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zheng R, Zhang S, Zhao P, Zeng H, Zou X. Report of cancer incidence and mortality in China, 2010. Ann Transl Med. 2014 Jul;2(7):61. doi: 10.3978/j.issn.2305-5839.2014.04.05. PMID 25333036
- [Background] Wagner M, Redaelli C, Lietz M, Seiler CA, Friess H, Buchler MW. Curative resection is the single most important factor determining outcome in patients with pancreatic adenocarcinoma. Br J Surg. 2004 May;91(5):586-94. doi: 10.1002/bjs.4484. PMID 15122610
- [Background] Willett CG, Czito BG, Bendell JC, Ryan DP. Locally advanced pancreatic cancer. J Clin Oncol. 2005 Jul 10;23(20):4538-44. doi: 10.1200/JCO.2005.23.911. PMID 16002845
- [Background] Iacobuzio-Donahue CA, Fu B, Yachida S, Luo M, Abe H, Henderson CM, Vilardell F, Wang Z, Keller JW, Banerjee P, Herman JM, Cameron JL, Yeo CJ, Halushka MK, Eshleman JR, Raben M, Klein AP, Hruban RH, Hidalgo M, Laheru D. DPC4 gene status of the primary carcinoma correlates with patterns of failure in patients with pancreatic cancer. J Clin Oncol. 2009 Apr 10;27(11):1806-13. doi: 10.1200/JCO.2008.17.7188. Epub 2009 Mar 9. PMID 19273710
- [Background] Koong AC, Le QT, Ho A, Fong B, Fisher G, Cho C, Ford J, Poen J, Gibbs IC, Mehta VK, Kee S, Trueblood W, Yang G, Bastidas JA. Phase I study of stereotactic radiosurgery in patients with locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1017-21. doi: 10.1016/j.ijrobp.2003.11.004. PMID 15001240
- [Background] Koong AC, Christofferson E, Le QT, Goodman KA, Ho A, Kuo T, Ford JM, Fisher GA, Greco R, Norton J, Yang GP. Phase II study to assess the efficacy of conventionally fractionated radiotherapy followed by a stereotactic radiosurgery boost in patients with locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):320-3. doi: 10.1016/j.ijrobp.2005.07.002. PMID 16168826
- [Background] Schellenberg D, Goodman KA, Lee F, Chang S, Kuo T, Ford JM, Fisher GA, Quon A, Desser TS, Norton J, Greco R, Yang GP, Koong AC. Gemcitabine chemotherapy and single-fraction stereotactic body radiotherapy for locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):678-86. doi: 10.1016/j.ijrobp.2008.01.051. Epub 2008 Apr 18. PMID 18395362
- [Background] Herman JM, Chang DT, Goodman KA, Dholakia AS, Raman SP, Hacker-Prietz A, Iacobuzio-Donahue CA, Griffith ME, Pawlik TM, Pai JS, O'Reilly E, Fisher GA, Wild AT, Rosati LM, Zheng L, Wolfgang CL, Laheru DA, Columbo LA, Sugar EA, Koong AC. Phase 2 multi-institutional trial evaluating gemcitabine and stereotactic body radiotherapy for patients with locally advanced unresectable pancreatic adenocarcinoma. Cancer. 2015 Apr 1;121(7):1128-37. doi: 10.1002/cncr.29161. Epub 2014 Dec 23. PMID 25538019
- [Background] Peretz T, Nori D, Hilaris B, Manolatos S, Linares L, Harrison L, Anderson LL, Fuks Z, Brennan MF. Treatment of primary unresectable carcinoma of the pancreas with I-125 implantation. Int J Radiat Oncol Biol Phys. 1989 Nov;17(5):931-5. doi: 10.1016/0360-3016(89)90138-7. PMID 2808054
- [Background] 王俊杰，黄毅，冉宝强．放射性粒子组织间种植治疗肿瘤临床应用的可行性IJ]． 中国微创外科杂志．2003．3：148．149．
- [Background] Zhang FJ, Wu PH, Zhao M, Huang JH, Fan WJ, Gu YK, Liu J, Zhang L, Lu MJ. [CT guided radioactive seed 125I implantation in treatment of pancreatic cancer]. Zhonghua Yi Xue Za Zhi. 2006 Jan 24;86(4):223-7. Chinese. PMID 16677499
- [Background] 王忠敏，陈克敏，金冶宁等.CT 引导下植入 125I 粒子放射性粒子治疗胰腺癌的疗效观 察[J].中国肿瘤临床，2009,36:65-69.
- [Background] 朱永强，陈俊英，郭剑锋.CT 引导下 125I 粒子植入治疗晚期胰腺癌的临床疗效分析[J]. 介入放射学杂志，2011,20（4）：283-286
- [Background] 盖宝东，舒振波，丁大勇等．125I放射性粒子治疗胰腺癌[J]．中国普外基础与临床杂 志．2007．14(5)：582-583．
- [Background] 熊炯忻，黄鹏，王春友．125I粒子组织间植入治疗局部进展期胰腺癌42例[J]．中国肿 瘤临床，2005．32(23)：1352一1355．
- [Background] 李振家，肖连祥，胰腺癌CT导引近距离放疗穿刺入路选择技术及策略[J]．当代医学． 2009．1 5(29)：543-546．
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415